CLINICAL TRIAL: NCT06737536
Title: A Single- and Multiple-ascending Dose Study to Investigate Safety, Tolerability and Pharmacokinetics of NNC0662-0419 in Participants Living With Overweight or Obesity
Brief Title: A First-in-human Research Study on How NNC0662-0419 Works in People Living With Overweight or Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: NN9662-7694; U1111-1304-7446 (Other: World Health Organization (WHO))
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: Single ascending dose (SAD) (Experimental): Participants will receive a single dose of any of the five different dose levels of NNC0662-0419 or matching placebo in a sequential manner with the dose increasing between cohorts.
  Interventions: Drug: NNC0662-0419; Other: Placebo (NNC0662-0419)
- Part B: Multiple ascending dose (MAD) (Experimental): Participants will receive NNC0662-0419 once-weekly for 4 weeks at any of the four different dose levels or matching placebo in a sequential manner with the dose increasing between cohorts.
  Interventions: Drug: NNC0662-0419; Other: Placebo (NNC0662-0419)

INTERVENTIONS:
Drug: NNC0662-0419 — Participants will receive NNC0662-0419 subcutaneous (s.c.) once weekly.
Other: Placebo (NNC0662-0419) — Participants will receive placebo matched to NNC0662-0419 s.c. once weekly.

SUMMARY:
This study is testing a new study medicine which may be used to treat people living with overweight or obesity. The purpose of the study is to see if the new study medicine is safe, how it works in human body and what human body does to the study medicine. Participants will either get the study medicine NNC0662-0419 or placebo (a "dummy" medicine without any active ingredients) given by study staff as an injection under participants skin. Which treatment participants will get is decided by chance. NNC0662-0419 is a new medicine, which cannot be prescribed by doctors. This is the first time the medicine is being given to humans. The study will last for about 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (sex at birth)
* Aged 19-55 years (both inclusive) at the time of signing the informed consent.
* Body mass index (BMI) between 27.0 and 39.9 kilogram per square meter (kg/m^2) (both inclusive) at screening. Overweight should be due to excess adipose tissue, as judged by the investigator.
* Considered eligible based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

* Known or suspected hypersensitivity to study intervention(s) or related products.
* Any disorder, unwillingness or inability which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol.
* 2nd or 3rd degree atrioventricular-block, prolongation of the QRS complex over 120 milliseconds (ms), or of the corrected QT interval by Fridericia (QTcF) calculation over 450 ms (females) or 430 ms (males), or any other clinically significant abnormal ECG results as judged by the investigator, at screening.
* Glycated haemoglobin (HbA1c) greater than or equal to (>=) 6.5 percent (%) (48 millimoles per mole [mmol/mol]) at screening.
* Calcitonin >= 50 nanogram per liter (ng/L) at screening

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2024-12-18 (Actual); Primary Completion 2025-07-26 (Actual); Study Completion 2025-07-26 (Actual)

PRIMARY OUTCOMES:
Part A: Number of treatment emergent adverse events (TEAE) | From timing of dosing on day 1 until completion of the end of study visit (up to 6 weeks)
  Number of events
Part B: Number of treatment-emergent adverse events (TEAE) | From timing of dosing on day 1 until completion of the end of study visit (up to 9 weeks)
  Number of events

SECONDARY OUTCOMES:
Part A: AUC; the area under the NNC0662-0419 plasma concentration-time curve | From pre-dose on day 1 until completion of the end of study visit (up to 6 weeks)
  measured in hour*nanomoles per liter (h*nmol/L)
Part A: Cmax; the maximum plasma concentration of NNC0662-0419 | From pre-dose on day 1 until completion of the end of study visit (up to 6 weeks)
  measured in nanomoles per liter(nmol/L)
Part B: AUC; the area under the NNC0662-0419 plasma concentration-time curve | From pre-dose on day 1 until completion of the end of study visit (up to 9 weeks)
  measured in h*nmol/L
Part B: Cmax; the maximum plasma concentration of NNC0662-0419 | From pre-dose on day 1 until completion of the end of study visit (up to 9 weeks)
  measured in nmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Celerion, Lincoln, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com